CLINICAL TRIAL: NCT02920073
Title: Intestinal Metagenome of Undernourished in Patients
Acronym: INT-METAVOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: INT-METAVOSA
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-08

CONDITIONS: Undernourished; Anorexia Nervosa
Keywords: Microbiota; anorexia nervosa; under nutrition; inpatients; enteral nutrition
MeSH Terms: conditions — Malnutrition; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this trial is to evaluate gut microbiota changes in undernourished patients with anorexia nervosa under enteral nutrition.

DETAILED DESCRIPTION:
This is a prospective, comparative, non-interventional study involving one clinical nutrition unit in France. Gut microbial will be evaluated with feces between patients and healthy volunteers.

Main investigations:

* Presence of gut microbial deviation compared to healthy volunteers;
* Presence of a significant statistical association between this deviation and metabolic disorders.

For each patient under the routine care a clinical examination and a blood sample will be done for standard biology report and nutrition. The age, gender, weight, height (for calculation of BMI), type of anorexia nervosa will be also collected with the pathological behavior associated (physical and intellectual hyperactivity, potomania, ongoing supplements drug taking including vitamins and trace elements). Eating and psychological disorders will be evaluated with EDI (eating disorder inventory) questionnaire.

Only the age, gender, height, weight (BMI), medical antecedents and ongoing treatment taking will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Anorexia nervosa as defined by DSM-5 (Diagnostic and Statistics Manual of Mental disorders
2. Undernutrition defined by BMI under 15
3. Age superior to 18
4. Patient hospitalised for undernutrition or seen in hospital day
5. Affiliation to the French social security regime or a similar regime
6. Patient signed informed consent

Healthy volunteers:

1. Age superior to 18
2. Normal weight (BMI 18.5 - 25)
3. Affiliation to the French social security regime or a similar regime
4. Patient signed informed consent

Exclusion Criteria:

Patients:

1. Taking antibiotics two month before hospitalization
2. Purge line with laxative abuse one month before hospitalization
3. Another disease may be associated to microbiota profile modification (diabetes, MICI or digestive organ pathology, metabolic disease)
4. Obesity prior to anorexia nervosa
5. Safeguard justice procedure

Healthy volunteers:

1. Metabolic anomaly
2. Recent weight change

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undernourished inpatients with anorexia nervosa under enteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change of the gut microbiota in undernourished inpatients with anorexia nervosa compared to healthy subjects. | 1 day

SECONDARY OUTCOMES:
Presence of a significant statistical association between this changes and metabolic troubles. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Hanachi-Guidoum, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Raymond Poincaré, Garches, France